CLINICAL TRIAL: NCT02372110
Title: Disentangling Anxiety Sensitivity and Anxiety-induced Physiological Stress Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Robert Josephs, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2015010023
Record Dates: First submitted 2015-02-12; First posted 2015-02-26 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Caffeine; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HPA, ANS stimulation (Experimental): Oral administration of 400mg caffeine and 20mg hydrocortisone will stimulate HPA axis and ANS activity, respectively
  Interventions: Drug: HPA, ANS stimulation
- Two cellulose placebo capsules (Placebo Comparator): two cellulose capsule filled with acidophilus powder will be administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HPA, ANS stimulation — Oral administration of Hydrocortisone will increase HPA axis activity. Oral administration of Caffeine will boost ANS activity
  Other Names: vivarin, cortef
  Arms: HPA, ANS stimulation
Drug: Placebo — Two cellulose placebo capsules filled with acidophilus powder will be administered to subjects who are randomly assigned to the placebo condition
  Other Names: fake pill
  Arms: Two cellulose placebo capsules

SUMMARY:
The proposed study aims to investigate experimentally anxiety sensitivity and physiologic sensations associated with anxiety using a paradigm combining hydrocortisone, caffeine, and a set of social stress challenges. Following informed consent, participants will be instructed to ingest either 400 milligrams of caffeine (an amount of caffeine roughly equivalent to that in two 8 oz. cups of brewed coffee from Starbucks), and 20 milligrams of hydrocortisone or two placebo capsules via stratified, random assignment. Physiologic and self-reported measures of stress and anxiety will be taken.

DETAILED DESCRIPTION:
Given the debilitating nature of anxiety disorders, a greater understanding of its etiology and the development of appropriate early interventions are critical. However, due to the mutually reinforcing nature of anxiety sensitivity (a key component of anxiety disorders) and physiological sensations associated with anxiety, no previous studies have examined these two variables separately in response to an acute stressor. The proposed study aims to investigate these two variables independently using a paradigm combining hydrocortisone, caffeine, and TSST.

It is hypothesized that when an individual's physiological stress responses (SNS and HPA axis) are enhanced, he or she will experience greater subjective stress and a lesser sense of mastery in response to an acute stressor (e.g., the TSST). In addition, anxiety sensitivity will moderate subjective ratings of stress and mastery, such that individuals high on anxiety sensitivity will rate the TSST as more subjectively stressful and their performance as less effectual compared to individuals low on anxiety sensitivity, due to greater vigilance of interoceptive responses and internal stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female participants will be required to pass the telephone-screening questionnaire. All eligible participants will be 18 years and older.

Exclusion Criteria:

* Full physiological exclusions include: abnormal electrocardiogram (i.e., arrhythmias), allergy to hydrocortisone or caffeine, anemia, cancer, chronic pain, compromised immune system (e.g., HIV), congestive heart failure, diabetes, diverticulitis, epilepsy, gastroesophageal reflux disease, gastrointestinal disease (e.g., bleeding), heart disease, hepatic impairment, herpes virus, high blood pressure or low blood pressure, high cholesterol, history of stroke, hypothyroidism, infection/fever in the last 7 days, kidney disease, liver disease (e.g., hepatitis), migraines/chronic headaches, myasthenia gravis, ocular herpes simplex virus, osteoporosis, peptic ulcer disease, renal impairment, respiratory disease (e.g., asthma), seizure disorder, skeletal muscle disease, spastic colon, strongyloides infection, surgeries within the last 6 weeks, systemic fungal infection, thyroid disease, tuberculosis/history of positive tuberculosis test, and ulcerative colitis.

Full medication exclusions include: ADHD medication, antibiotics in the last 7 days, antidepressants, antiplatelet drugs, anxiolytics, bipolar disorder medication, blood pressure medication, blood thinners, bronchodilators, drugs for allergies, drugs to treat hormonal disorders, estrogen, insulin, live vaccinations in the last 7 days, long-lasting decongestants, pain killers (i.e., NSAIDS: aspirin or ibuprofen), sleeping pills, statins (i.e., to lower cholesterol), steroids.

Full psychological exclusions include current or previous diagnosis of major depression, posttraumatic stress disorder, specific phobia, anxiety disorders, or any other psychiatric condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Heart Rate | 180 minutes
  continuous heart rate monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Josephs, Ph.D, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States